CLINICAL TRIAL: NCT06144021
Title: 12 Weeks, Randomized, Double-blind, Placebo-controlled Trial on the Efficacy and Safety of Kefir Whey Postbiotics
Brief Title: Efficacy and Safety of Kefir Whey Postbiotics
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hanyang University Seoul Hospital (Other)
Collaborators: Ottogi Ham Taiho Foundation (Unknown); Hanyang University (Other)
Responsible Party: Principal Investigator, Jun Yup Kim, Clinical Assistant Professor, Hanyang University Seoul Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: HYUH 2023-07-059-008
Record Dates: First submitted 2023-11-09; First posted 2023-11-22 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Sarcopenia
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Intervention Model Description: Double-blind randomized controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: * During the trial period, neither the researcher nor the research subjects know the randomization information of the research subjects. In principle, the randomization code is maintained and stored by the researcher.
  * In general, double blinding should not be lifted until all research subjects have completed the test and the data is locked. However, in the case of an emergency such as a health problem of a research subject during intervention, double blinding may be lifted at the discretion of the researcher. In this case, the research person must contact the principal investigator as quickly as possible.
  * The date, time, and reason for lifting double blinding must be documented in an appropriate location in the case record and supporting documents. A copy of the double-blind code release confirmation document received from the principal investigator must be kept in the supporting documents.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kefir Postbiotics Group (Experimental): * 30 healthy adult participants
  * Appearance and formulation: Yellow powder/capsule with unique flavor and no off-flavor
  * Period of use: 12 months
  * Storage method: Store at room temperature
  * Manufacturing method: The whey postbiotics derived from kefir lactic acid bacteria used in the test food are produced in the laboratory at Hanyang University, and additional ingredients are purchased from finished products. Laboratory collects the ingredients and delivers them to the manufacturer, Neo Natural, to manufacture them so that there are no differences in properties and formulations.
  Interventions: Dietary Supplement: Whey postbiotics derived from kefir lactic acid bacteria
- Control Group (Placebo Comparator): * 30 healthy adult participants
  * Appearance and formulation: Yellow powder/capsule with unique flavor and no off-flavor
  * Period of use: 12 months
  * Storage method: Store at room temperature
  * Manufacturing method: The same product without whey postbiotics.
  Interventions: Dietary Supplement: Placebo powder

INTERVENTIONS:
Dietary Supplement: Whey postbiotics derived from kefir lactic acid bacteria — Kefir (alcoholic fermented dairy product made by fermenting cow, goat, or sheep milk) whey derived from lactic acid bacteria postbiotics
  Arms: Kefir Postbiotics Group
Dietary Supplement: Placebo powder — A powder product including Flavor, Calcium carbonate, Lactose, Maltodextrin, Sugar, Carboxy methyl cellulose. This cannot be distinguished from the postbiotics by inspection.
  Arms: Control Group

SUMMARY:
Research staff conduct screening tests only on applicants who provide written consent and select research subjects who meet the selection criteria. Study subjects will visit for the first time within 4 weeks from the screening visit to reexamine the suitability of the study subject selection/exclusion criteria and then be enrolled in the human application test. The participants will be randomly assigned to the kefir lactic acid bacteria-derived whey post-biotics group and the placebo group for the first time. Complete the baseline evaluation by the date of visit. Afterwards, the participants will consume whey postbiotics derived from kefir lactic acid bacteria and a placebo product twice a day, 3g per time, for 12 weeks, and visit the institution a total of four times to perform a grip strength test, DXA, etc. This survey will be conducted at Hanyang University Hospital. Research staff may conduct follow-up observations of study subjects as needed after final consumption of the kefir lactic acid bacteria-derived whey postbiotic group and placebo products or after early termination.

DETAILED DESCRIPTION:
Purpose: Kefir (alcoholic fermented dairy product made by fermenting cow's milk, goat's milk, or sheep's milk) to determine the effect of 12 weeks of human consumption of whey postbiotics derived from lactic acid bacteria in improving muscle strength and intestinal microbiome in elderly people compared with placebo intake.

-Primary objective: To evaluate the effectiveness of whey postbiotics derived from kefir lactic acid bacteria compared to placebo intake through the results of the grip strength test for both hands.

-Secondary objective: To evaluate the effectiveness and safety of whey postbiotics derived from kefir lactobacilli for muscle strength improvement as assessed by dual energy x-ray absorptiometry (DXA), adipokines, myokines, and cytokines compared with placebo intake. The investigators aim to analyze the differences in the intestinal microbiome compared to placebo intake through fecal collection and NGS (Next Generation Sequencing).

Experimental product: Kefir lactic acid bacteria-derived whey postbiotics (oral intake of 6g per day (3g twice per day))

Control product: Flavor 2.7%, Calcium carbonate 13.8%, Lactose 41.3%, Maltodextrin 10.3%, Sugar 31.23%, Carboxy methyl cellulose 0.67% (oral intake of 6g per day (3g twice per day))

Number of subjects: In this human application test, in order to calculate the number of study subjects, the investigators referred to previous studies and calculated the lean mass gain (kg) of 3.3 ± 1.5 kg (mean ± SD) after consuming whey postbiotics derived from kefir lactic acid bacteria for 12 weeks. In the placebo group, it was assumed to be 1.8 ± 1.6 kg.

* The statistical hypothesis test of the evaluation variable is a two-sided test.

  * The significance level is 5%. ③ The test power is maintained at 90% and the type 2 error is set at 0.2. ④ The ratio between the test group and the control group is divided at 1:1.

    * The calculation of the number of subjects referred to existing research, and a T-test was performed using the G power program to use the mean of the statistical difference in muscle strength improvement between the two groups divided according to the intake of whey postbiotics derived from kefir lactic acid bacteria as the mean (test power) (1-β)=0.9, significance level (α)=0.05, effect size (ES)=0.97 (Cohen's d)). The total number of research subjects required for human application testing calculated through this is 48. Here, the investigators plan to recruit a total of 60 research subjects, assuming a dropout rate of 20%.

ELIGIBILITY:
Inclusion Criteria:

1. Adult men and women aged 40 years or older at the time of screening test
2. Adult men and women with a Charlson Comorbidity Index (CCI) score of 0 at the time of screening
3. Adult men and women with skeletal muscle mass less than 110% of the standard as measured by BIA (bioelectrical impedence analysis) at the time of screening test

Exclusion Criteria:

1. Those with significant hypersensitivity to melon gourd, whey, or lactic acid bacteria ingredients
2. Those who participated in other human application tests, diet, or exercise programs within 3 months before the screening test
3. Persons with clinically significant acute or chronic cardiovascular, diabetes, endocrine, immune, respiratory, hepatobiliary, renal and urinary, neuropsychiatric, or gastrointestinal diseases requiring treatment.
4. Those who show the following results in blood or urine tests:

   * AST, ALT > 1.5 times the upper limit of the reference range
   * Serum Creatinine > 1.4 mg/dL
   * Fasting blood sugar > 126mg/dL
5. If there is 2+ or more proteinuria
6. Persons taking medication for psychiatric illness (excluding cases of intermittent medication due to sleep disorders)
7. Those who consumed pro- or prebiotics within 1 month before the screening test
8. Those who have taken protein supplements regularly for more than 3 months within 6 months before the screening test
9. Those who received other investigational drugs within 1 month before the screening test
10. Those who received antibiotics within 2 months before the screening test
11. Those who are currently controlling their diet for disease management purposes
12. Those with a history of gastrointestinal resection (excluding the appendix)
13. Those who are performing or plan to perform regular resistance exercise
14. People with vegetarian beliefs
15. People with food allergies or restricted foods
16. Persons with a history of diagnosed gastrointestinal disease (ex. ulcerative colitis, Crohn's disease, gastroparesis, peptic ulcer disease, cancer, celiac disease, short bowel, and ileostomy)
17. Those taking constipation or diarrhea medication
18. Those who currently smoke
19. Those whose BMI exceeds 30kg/m2 at the time of screening test
20. Those who plan to control their weight within 6 months after screening
21. Those who are likely to be uncooperative in this test or those who are determined by the researcher to be unable to proceed with the test

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-12-15 (Actual); Primary Completion 2024-10-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Grip strength test for both hands | 1) Day 0, 2) end of 12 weeks
  Handgrip strength should be measured using the JAMAR grip dynamometer (Jamar, Plus+ Digital Hand Dynamometer, Preferred, USA). While the research subject is sitting, the grip strength of both hands is measured three times each, and the average value is taken as the representative value. The unit of grip strength is kg.
Dual energy xray absorptiometry | 1) Day 0, 2) end of 12 weeks
  Dexa imaging measures the whole body, lean mass, body fat mass, and bone mineral content using Hanyang University Hospital's DXA (Discovery W DEXA) equipment after fasting for more than 8 hours. Measurements will be taken with the study subject standing upright, rotating both feet inward about 15 degrees, and placing both hands next to the waist. Here, the investigators will measure skeletal muscle mass (SMM, kg) by subtracting bone mineral content (BMC) from lean body mass. And the SMM and the height (m) will be combined to report skeletal muscle mass index (SMMI) in kg/m^2 unit.

SECONDARY OUTCOMES:
Biomarkers from blood | 1) Day 0, 2) end of 12 weeks
  All in ng/mL
  : 1) adipokines (leptin, adiponectin) 2) myokines (myostatin, irisin) 3) lipid analysis (TG, T-C, HDL-C, LDL-C) 4) cytokines (CRP, IL-2, IL-6, IL-1β, TNF-α, IGF-1)
Confirmation of intestinal microorganisms | 1) Day 0, 2) end of 12 weeks
  Stool collection is collected directly by the research subject 1 day before (24 hours) before the start of consumption of whey postbiotics derived from kefir lactic acid bacteria and after the last intake, and stored at a frozen temperature (-20℃ or lower) until the first and third visits. do. Research staff collect stool samples, store them frozen (-70°C), and then perform next-generation sequencing (NGS analysis).

CONTACTS AND LOCATIONS:
Locations (1):
- Hanyang University Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No